CLINICAL TRIAL: NCT04816487
Title: Effect of Glutathione vs Potassium Iodide in Reducing Silver Diamine Flouride Staining When Used in Treatment of Primary Carious Teeth
Brief Title: Effect of Glutathione vs KI in Reducing SDF Staining When Used in Treatment of Primary Carious Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Abdulaziz Hifni, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Reducing discoloration of SDF
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Discoloration, Tooth
MeSH Terms: conditions — Tooth Discoloration | interventions — Potassium Iodide; Glutathione

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silver Diamine Flouride (Active Comparator): Discoloration of primary carious teeth treated by SDF
  Interventions: Drug: Potassium Iodide or Glutathione
- Glutathione (Experimental): Discoloration rate of primary carious teeth treated by SDF + Glutathione
  Interventions: Drug: Potassium Iodide or Glutathione
- Potassium iodide (Experimental): Discoloration rate of primary carious teeth treated by SDF + KI
  Interventions: Drug: Potassium Iodide or Glutathione

INTERVENTIONS:
Drug: Potassium Iodide or Glutathione — Patient will receive either Glutathione or Potassium iodide

SUMMARY:
Although black staining is considered a drawback that is clinically observed following SDF application and is the main primary barrier for its use clinically . Child's behaviour and cooperation cannot be controlled at a young age or in special health care needs cases. Therefore, the best treatment modality will always be a simple, fast and painless procedure and SDF is the best solution for those cases. Discolouration caused researchers to search for a solution that will reduce or prevent discolouration using KI and GSH. A systematic review was conducted in-vitro, and it showed the use of SDF with KI had reduced stains markedly, potential advantages of minimal staining might be advantageous, along a short period. However, studies with long-term follow-up would be required to provide evidence-based guidelines for using SDF and KI formulations in routine clinical practice

DETAILED DESCRIPTION:
Early childhood caries (ECC) has been increasing worldwide and became a significant health problem. ECC is a multifactorial disease result from the interaction of different factors as cariogenic microorganisms, exposure to fermentable carbohydrates through inappropriate feeding habits. It affects teeth that are less susceptible to caries. The management of ECC is expensive, often requiring extensive restorative treatment such as the drill and fill technique and extraction of teeth at an early age. Nowadays, non-invasive treatment for arresting untreated dental caries is becoming urgently needed.

Silver diamine fluoride (SDF) treatment offers an alternative non-invasive treatment for caries as it arrests caries progression. S.D.F. is a colourless agent in the form of liquid with an alkaline PH of 10 it contains 24.4% to 28.8% (weight/volume) silver and 5.0 to 5.9% fluoride .. SDF is inexpensive treatment, and its ease of the application makes it a durable treatment option in dental clinics. Arresting active caries is an essential treatment modality and requires training by all dental auxiliaries.

The major drawback to SDF treatment has been its black stain and discolouration, which has limited its use. The precipitation of silver by-products in the dental tissues results in black staining, which can be discouraging and limits its use in visible areas. SDF also temporarily stains skin and gingiva, requiring them to be handled carefully to avoid contact with these tissues. To overcome the staining, SDF researchers investigated applying a saturated solution of potassium iodide (10% weight % KI) and studied the effect of glutathione (GSH) biomolecule on reducing of enamel and dentin discolouration.

Potassium iodide (KI) is used as a nutritional supplement. A supersaturated solution of KI is used in managing the discolouration problem of the carious lesion without affecting its caries arresting effect. It reduces the staining caused by the SDF as silver ions from the SDF solution reacts with the iodide ions present in KI solution, which results in the formation of silver iodide.

Glutathione (GSH) is a tri-peptide biomolecule, and it is considered one of the best with silver as it contains a thiol group (-SH) which has a high affinity for adsorption onto metal surfaces . GSH also forms a coat around silver particles, decreasing the aggregation of silver particles and controlling the rate of silver ion release (Homeostasis) , which reduces the discolouration of an SDF-coated tooth over time. This study was conducted to compare the effect of glutathione (GSH) versus Potassium iodide (KI) in reducing the SDF staining effect in carious primary teeth.

ELIGIBILITY:
Inclusion Criteria:

-

Children:

* Aged 3 to 5 years, in good general health and medically free.
* The parents provided written informed consent.
* Medically free

Teeth:

* Carious primary teeth
* Restorable teeth.
* Teeth are not pulpally involved

Exclusion Criteria:

* Children:

  * with a history of allergy to silver
  * Unable to attend follow-up visits.
  * Refusal of participation.

Teeth:

* Previously restored teeth.
* Periapical swelling and tenderness in this area.
* With mobility.
* With spontaneous pain.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Colour assessment | 6 months
  Using Vita easy shade ( continuous) ΔE

SECONDARY OUTCOMES:
Parenteral satisfaction | 6 months
  Direct using questionnaires Binary (Yes/No)
3-Side effects Gum swelling Gum bleaching Tooth or gum pain Nausea 3-Side effects Gum swelling Gum bleaching Tooth or gum pain Nausea 3-Side effects Gum swelling Gum bleaching Tooth or gum pain Nausea Side effects | 6 months
  Direct using questionnaires Binary (Yes/No)